CLINICAL TRIAL: NCT05524207
Title: A Controlled Clinical Study of Carotid Artery Stent Implantation in the Treatment of Vulnerable Plaque
Brief Title: Carotid Artery Stent Implantation in the Treatment of Vulnerable Plaque
Acronym: CASTLE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Principal Investigator, Keqiang Zhao, Attending Doctor, Beijing Tsinghua Chang Gung Hospital
Other Study IDs: 20220816
Record Dates: First submitted 2022-08-30; First posted 2022-09-01 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Carotid Artery Plaque; Carotid Stenosis; Stent Embolisation
Keywords: carotid artery stenosis; vulnerable plague; carotid stenting
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vulnerable plaque group: Patients with preoperative contrast-enhanced intra-plaque contrast agent were classified as vulnerable plaque group
  Interventions: Procedure: carotid artery stenting
- Stable plaque group: The patients with no contrast agent enhancement in the plaque showed preoperative contrast-enhanced ultrasound were classified as stable plaque group
  Interventions: Procedure: carotid artery stenting

INTERVENTIONS:
Procedure: carotid artery stenting — Implantation of stents at the site of carotid artery stenosis for the treatment of carotid plaque with severe stenosis

SUMMARY:
To investigate the efficacy and safety of carotid stenting for vulnerable carotid plaques. All patients with carotid artery stenosis underwent carotid arterial contrast-enhanced ultrasonography before operation. According to the examination results, they were divided into two groups: vulnerable plaque group and stable plaque group. The incidence of perioperative stroke events in the two groups was compared. The incidence of stroke events in the two groups within 1 year was compared.

DETAILED DESCRIPTION:
1. To enroll 100 cases of patients suffering from carotid artery stenosis。the investigators perform contrast enhanced ultrasound on patients for identifying the vulnerable plagues
2. The investigators divide patients into the stable group and the vulnerable group based on the results of CEUS inspection.
3. All patients undergo carotid stent. To analysis the incidence of postoperative complications such as stroke and mortality within 30 days and to compare the differences between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* The patients with ischemic symptom whose carotid stenosis were more than 50%
* The patients without ischemic symptom whose carotid stenosis were more than 70%

Exclusion Criteria:

* • Confirmed with severe intracranial vascular lesions

  * Suffering from the large area cerebral infarction or critical stroke sequela
  * Restenosis after CEA or CAS
  * Suffering from severe coronary heart disease, respiratory failure,the hypertension difficult to controled
  * Patients with malignant tumor or expected life < 2 years

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the patients suffering from carotid artery stenosis
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Perioperative 30-day stroke rate | 30 days
  To determine whether there is a new cerebral infarction by postoperative re-examination of brain MRI and preoperative brain MRI

SECONDARY OUTCOMES:
1-year stroke rate after surgery | 1 year
  Stroke rate in ipsilateral carotid artery blood supply area within 1 year after operation

CONTACTS AND LOCATIONS:
Overall Officials: sifan yang, Study Director — Beijing Tsinghua Chang Gung Hospital
Locations (1):
- Beijing Tsinghua Chang Gung Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No